CLINICAL TRIAL: NCT05328232
Title: Effects of Olive Oil Use on The Healing of Diaper Rash
Brief Title: The Effect Of Olive Oil on Diaper Rash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Nejla Canbulat Şahiner, Prof. Dr., Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/09
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Diaper Rash; Olive Oil
MeSH Terms: conditions — Diaper Rash | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil (Experimental)
  Interventions: Other: Olive oil
- Routine care (No Intervention)

INTERVENTIONS:
Other: Olive oil — The parents of the babies included in the experimental group were asked to fill in the questionnaires. The infant's skin condition was assessed using the Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants. Each time the diaper was changed, the diaper area was cleaned with water and cotton wool and dried, 1-2 cc of natural extra virgin olive oil was applied, and the new diaper was fastened. At the end of each day, the diaper area was evaluated by the researcher and a nurse by using the Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants.
  Arms: Olive oil

SUMMARY:
Objective: Diaper rash is an irritating, common skin problem in newborns and young children and occurs in the skin rubbed by wet diapers and in the armpits due to heat, moisture and irritation. This experimental study was planned to investigate the effect of olive oil use on the healing of diaper rash in infants with first-degree diaper rash undergoing treatment in an infant ward.

Methods: The study conducted between September 2020 and December 2020 included 37 infants aged 0-24 months who were treated for any reason in the Infant Clinic of a medical school and had first-degree rash. The infants in the experimental and control groups were "treated with olive oil and X brand cream" respectively. The X brand cream and the effects of olive oil and X brand cream use on the improvement of diaper rash were compared.

ELIGIBILITY:
Inclusion Criteria:

* Having a first-degree diaper rash
* Being 0-24 months old
* Having the family's consent indicating that they allow their child to be included in the study

Exclusion Criteria:

* The baby's having anorectal congenital anomaly
* The baby's having an obstacle to the application of olive oil (allergy, etc.)
* Having a second-degree or third-degree rash

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the scores obtained from the Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants by the Experimental and Control Groups. | October-November 2020 (two months)
  comparison of the scores obtained from the Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants by the Experimental and Control Groups

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adalat S, Wall D, Goodyear H. Diaper dermatitis-frequency and contributory factors in hospital attending children. Pediatr Dermatol. 2007 Sep-Oct;24(5):483-8. doi: 10.1111/j.1525-1470.2007.00499.x. PMID: 17958792. 2. Atherton DJ. The Aetiology and Management of Irritan Diaper Dermatitis. European Academy of Dermatology and Venereology, 2001;15:1-4. 3. Al-Waili N.S. Clinical and Mycological Benefits of Topical Application of Honey, Olive oil and Beeswax in Diaper Dermatitis. Clinical Microbiology and Infection, 2005;11(2): 141-163. 4. Arısoy A, Canbulat N, Ayhan A. Karaman İlindeki Annelerin Bebeklerinin Bakımında Uyguladıkları Geleneksel Yöntemler. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 2014;17(1): 23-32. 5. Buckley BS, Mantaring JB, Dofitas RB, Lapitan MC, Monteagudo A. A New Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants, Development and Validation. Pediatric Dermatology, 2016,33(6):632-639. 6. Danby SG, Alenezi T, Sultan A, Lavender T, Chittock J, Brown K, Cork MJ. Effect of Olive and Sunflower Seed Oil on the Adult Skin Barrier, İmplications for Neonatal Skin Care. Pediatric Dermatology, 2013;30(1):42-50. 7. Duffy LJ, Ferguson MR, Darmstadt LG. Opportunities for Improving, Adapting and Introducing Emollient Therapy and Improved Newborn Skin Care Practices in Africa. Journal of Tropical Pediatrics. 2012;58(2): 88-95. 8. Felter SP, Carr AN, Zhu T, Kirsch T, Niu G. Safety Evaluation for İngredients Used in Baby Care Products: Consideration of Diaper Rash. Regulatory Toxicology and Pharmacology, 2017;90:214-221. 9. Fölster-Holst R. Differential Diagnoses of Diaper Dermatitis. Pediatric Dermatology, 2018;35:10-18. 10. Gözen D, Çağlar S, Bayraktar S, Atıcı F. Diaper Dermatitis Care of Newborns Human Breast Milk or Barrier Cream. Journal of Clinical Nursing, 2013;23(3-4):515-523. 11. Gupta AK, Skinner AR. Management of Diaper Dermatitis. Int J Dermatol, 2004;43: 830-834. 12. Kenner C, Lott JW, Flandermeyer A. A Comprehensive Neonatal Nursing. WB Saunders, Philadelphia, 1998;2:67-58. 13. Keskin E. Bebeklerde Komplike Olmayan Bez Dermatiti Şiddet Değerlendirme Ölçeğinin Geçerlik ve Güvenirliğinin İncelenmesi. Yüksek Lisans Tezi, Ege Üniversitesi Sağlık Bilimleri Enstitüsü, 2019, İzmir. 14. Kohlendorfer-Kiechl U, Berger C. Inzinger R. The Effect of Daily Treatment with an Olive Oil/Lanolin Emollient on Skin Integrity in Preterm Infants: A Randomized Controlled Trial. Pediatric Dermatology. 2008;25(2): 174178. 15. Kirlek F. Erken Pospartum Dönemde Meme Başı Ağrısı ve Çatlaklarının Önlenmesinde Anne Sütü ve Zeytinyağının Etkisi. Yüksek Lisans Tezi, Adnan Menderes Üniversitesi Sağlık Bilimleri Enstitüsü, 2010, Aydın. 16. Lupiáñez-Pérez I, Morilla-Herrera JC, Ginel-Mendoza L, Martín-Santos FJ, Navarro-Moya FJ, Sepúlveda-Guerra RP, Morales-Asencio JM. Effectiveness of Olive Oil for the Prevention of Pressure Ulcers Caused in İmmobilized Patients Within the Scope of Primary Health Care, Study Protocol for A Randomized Controlled Trial. Trials, 2013;14(1):1-7. 17. Mandleco BL. Theoretical Approaches to the Growth and Development of Children. In Pediatric Nursing Caring for Children and Their Families. (Eds). Micki L. Potts. United States of America. Delmar Thomsan Learning. 2002. 18. Nield LS, Kamat D. Prevention, Diagnosis and Management of Diaper Dermatitis. Clin Pediatr, 2007;46:480-486. 19. Önder M, Adışen E, Velagiç Z. Diaper Dermatit. Çocuk Sağlığı ve Hastalıkları Dergisi, 2007;50:129-135. 20. Panahi Y, Sharif MR, Sharif A, Beiraghdar F, Zahiri Z, Amirchoopani G, Sahebkar A. A Randomized Comparative Trial on the Therapeutic Efficacy of Topical Aloe Vera and Calendula Officinalis on Diaper Dermatitis in Children. The Scientific World Journal, 2012;20(12):1-5. 21. Pingvini S, Shahsavari S, Gazerani F, Abdolkavand S. Topical Use of Human Breast Milk for Diaper Rash in İnfants. Middle East Journal of Nursing, 2009;3:27-30. 22. Prasad HRY, Srivastava P, Verma KK. Diaper Dermatitis an Overview. The Indian Journal of Pediatrics, 2003;70(8):635-637. 23. Salam AR, Das KJ, Darmstadt LG, Bhutta AZ. Emollient Therapy for Preterm Newborn Infants-Evidence From the Developing World. BMC Public Health. 2013;13(3): 31-37. 24. Scheinfeld N. Diaper dermatitis. American journal of clinical dermatology, 2005;6(5): 273-281. 25. Sharifi-Heris Z, Amiri-Farahani L, Haghani H, Abdoli-Oskouee S, Hasanpoor-Azghady S. Comparison the Effects of Topical Application of Olive and Calendula Ointments on Children's Diaper Dermatitis. A Triple-blind Randomized Clinical Trial. Wiley Dermatology Therap, 2018;10(11):1-7. 26. Šikić Pogačar M, Maver U, Marčun Varda N, Mičetić-Turk D. Diagnosis and Management of Diaper Dermatitis in İnfants with Emphasis on Skin Microbiota in the Diaper Area. International Journal of Dermatology, 2018;57(3):265-275.